CLINICAL TRIAL: NCT01461226
Title: Adolescent Obesity: What Determines Vascular Endothelial Dysfunction And Is The Process Reversible?
Brief Title: Endothelial Dysfunction in Obese Children
Acronym: EDOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Zeepreventorium (Other)
Responsible Party: Principal Investigator, Luc Bruyndonckx, Principal Investigator, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC 11/11/100
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Atherosclerosis
Keywords: overweight; cardiovascular risk factors; exercise training; endothelial function; endothelium; endothelial progenitor cells
MeSH Terms: conditions — Obesity; Atherosclerosis; Overweight | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): Individualized and progressively increased supervised aerobic exercise program on a daily base (3-4hours per day, hypocaloric diet and psychological guidance
  Interventions: Behavioral: Exercise training
- Usual Care (Other): Nutritional assessment and dietary advice by general practitioner, promotion of sports activities
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Exercise training — Individualized and progressively increased supervised aerobic exercise program on a daily base (3-4hours per day, hypocaloric diet and psychological guidance
  Arms: Exercise training
Behavioral: Usual care — Nutritional assessment and dietary advice by general practitioner, promotion of sports activities
  Arms: Usual Care

SUMMARY:
The purpose of this study is to objectify the effect of diet and exercise on early markers of atherosclerosis in obese children.

DETAILED DESCRIPTION:
The favorable responses of combined treatment strategies, consisting of exercise training and proper diet change, for childhood and adolescent obesity on vascular health are poorly understood. The overall objective of this research project is to investigate the underlying pathophysiological mechanisms that mediate these beneficial effects.

Particularly, the following aims are set forth:

1. To establish the effect of a combined lifestyle intervention, i.e. an individualized exercise training and caloric restriction program, on vascular function (primary endpoint) and structure in a substantial population of obese adolescents.
2. To characterize causal pathways between obesity and endothelial dysfunction with focus on classical risk factors, oxidative and inflammatory stress, metabolic adaptations, bone marrow derived progenitor cells, and blood microparticles.

This research knowledge will be instrumental for risk stratification and clinical management aimed to improve endothelial function by limiting damage and reinforcing regenerative mechanisms in obese adolescents.

ELIGIBILITY:
Inclusion Criteria: Children with severe obesity

* Younger than 16 yrs: BMI ≥97th sex and age specific BMI-percentile
* Older than 16 yrs: BMI ≥35 kg/m²

Exclusion Criteria:

* Acute or chronic inflammatory process, use of non-steroidal anti- inflammatory drugs or immunosuppressive drugs. (including inhalation corticosteroids).
* Structural heart disease or other cardiac diseases.
* Active malignant hematological disease

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viviane M Conraads, M.D., PhD, Principal Investigator — Dienst Cardiale Revalidatie, Cardiologie, Universitair Ziekenhuis Antwerpen
Locations (3):
- Belgium (3):
  - Zeepreventorium, De Haan
  - Dienst Cardiale Revalidatie, Cardiologie, Universitair Ziekenhuis Antwerpen, Edegem
  - Dienst Pediatrie, Universitair Ziekenhuis Antwerpen, Edegem

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Training | Usual Care
Started | 33 | 28
Completed | 27 | 21
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Training | Usual Care | Total
Number analyzed (Participants) | 33 | 28 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 28 | 61
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.5) | 15 (1.2) | 15 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 9 | 6 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m²] | 36.44 (4.82) | 36.72 (5.83) | 36.58 (5.33)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Reactive Hyperemia Index at 5 and 10 Months
Description: Reactive Hyperemia Index as assessed using endoPAT (R) is used as a marker for endothelial function
Time Frame: Baseline - 5 months - 10 months
Population: this was an intention to treat analysis. Some participants ended the treatment.
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Exercise Training | Usual Care
Number analyzed (Participants) | 33 | 28
arbitrary units
  10 months: number analyzed (Participants) | 27 | 21
  10 months | 1.9 [1.5 to 3] | 1.5 [1.3 to 1.7]
  5 months: number analyzed (Participants) | 29 | 21
  5 months | 2.01 [1.58 to 2.50] | 1.55 [1.4 to 2.19]
  baseline | 1.48 [1.26 to 2.01] | 1.42 [1.24 to 1.84]
Statistical Analysis 1: Comparison: Exercise Training vs Usual Care; Test type: Other — Mixed models analysis; p < 0.05, Mixed Models Analysis; mixed models = 0.04
Statistical Analysis 2: Comparison: Exercise Training vs Usual Care; Test type: Other; p = 0.64, Mixed Models Analysis — Baseline difference between groups; mixed models = 0.24
Statistical Analysis 3: Comparison: Exercise Training vs Usual Care; Test type: Other — Mixed models; p = 0.60, Mixed Models Analysis; Slope = 0.27
Statistical Analysis 4: Comparison: Exercise Training vs Usual Care; change after 10 months between groups; Test type: Other — mixed models; p = 0.04, Mixed Models Analysis; mixed models = 4.2

2. Secondary Outcome: Change From Baseline in Exercise Capacity at 5 and 10 Months
Description: Exercise capacity will be assessed using bicycle ergometry at baseline and at 5 and 10 Months
Time Frame: Baseline - 5 months - 10 months
Population: this an intention to treat analysis. Some participants ended the treatment
Measure: Median (Inter-Quartile Range); unit: watt
Arm/Group | Exercise Training | Usual Care
Number analyzed (Participants) | 33 | 28
watt
  baseline | 150 [130 to 170] | 150 [130 to 170]
  5 months: number analyzed (Participants) | 29 | 21
  5 months | 170 [130 to 210] | 150 [130 to 170]
  10 months: number analyzed (Participants) | 27 | 21
  10 months | 170 [150 to 210] | 130 [130 to 170]

3. Secondary Outcome: Change From Baseline in Body Mass Index and Body Composition at 5 and 10 Months
Description: Weight and Length will be assessed to calculate Body Mass Index(BMI) at baseline and after 5 and 10 months
Time Frame: Baseline - 5 months - 10 months
Population: this is an intention to treat analysis. Some participants ended treatment
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Exercise Training | Usual Care
Number analyzed (Participants) | 33 | 28
kg/m²
  baseline | 36.44 (4.82) | 36.72 (5.83)
  5 months: number analyzed (Participants) | 29 | 21
  5 months | 30.07 (3.85) | 38.40 (5.62)
  10 months: number analyzed (Participants) | 27 | 21
  10 months | 27.39 (3.57) | 39.10 (5.26)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Exercise Training | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/28
Other Adverse Events (participants affected / at risk) | 0/33 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No